CLINICAL TRIAL: NCT06365957
Title: Acute Changes in Cardiometabolic and Neurocognitive Outcomes in Response to Exercise Combined With Ketone Ester Supplement in Overweight/Obese Adults
Brief Title: Acute Effects of Exercise Combined With Ketone Ester Supplement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BSERE24-APP001-FED
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity; Cognitive Change; Ketoses, Metabolic
Keywords: Overweight; Obesity; Exercise; Nutrients; Neurocognition; Metabolism
MeSH Terms: conditions — Overweight; Obesity; Ketosis; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- High-intensity interval exercise (HIIE)-Ketone Supplementation (KT) condition (Experimental): High-intensity interval exercise (HIIE) with ketone supplements [R-1,3-butanediol; San Francisco].
  Interventions: Other: Ketone monoester supplementation; Other: High-intensity interval exercise
- MICE-KT condition (Experimental): moderate-intensity continuous exercise (MICE) with ketone supplements.
  Interventions: Other: Ketone monoester supplementation; Other: Moderate-intensity continuous exercise
- Nonexercise (NE)-KT condition (Experimental): Non-exercise with ketone supplements.
  Interventions: Other: Ketone monoester supplementation
- HIIE-Placebo (PLA) condition (Experimental): HIIE with taste-matched placebo
  Interventions: Other: High-intensity interval exercise; Other: Placebo
- MICE-PLA condition (Experimental): MICE with taste-matched placebo
  Interventions: Other: Moderate-intensity continuous exercise; Other: Placebo
- NE-PLA condition (Experimental): Non-exercise with taste-matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ketone monoester supplementation — Exogenous ketones are a class of ketone bodies that are ingested using nutritional supplements or foods. This class of ketone bodies refers to the three water-soluble ketones (acetoacetate, β-hydroxybutyrate, and acetone).
  Arms: High-intensity interval exercise (HIIE)-Ketone Supplementation (KT) condition; MICE-KT condition; Nonexercise (NE)-KT condition
Other: High-intensity interval exercise — High-intensity interval exercise is a type of interval training exercise. It incorporates several rounds that alternate between several minutes of high-intensity movements to significantly increase the heart rate to at least 80% of one's maximum heart rate, followed by short periods of lower-intensity movements. The exercise will be conducted on a computer-monitored cycle ergometer.
  Arms: HIIE-Placebo (PLA) condition; High-intensity interval exercise (HIIE)-Ketone Supplementation (KT) condition
Other: Moderate-intensity continuous exercise — Moderate-intensity continuous exercise generally consists of 30-60 min of aerobic exercise at 64-76% peak heart rate, while interval training involves more intense bouts interspersed by recovery periods. The exercise will be conducted on a computer-monitored cycle ergometer.
  Arms: MICE-KT condition; MICE-PLA condition
Other: Placebo — The placebo will be the taste-matched water.
  Arms: HIIE-Placebo (PLA) condition; MICE-PLA condition; NE-PLA condition

SUMMARY:
To examine the acute changes in cardiometabolic and neurocognitive outcomes in response to exercise combined with ketone ester supplement in overweight/obese adults.

DETAILED DESCRIPTION:
The prevalence of excess body weight and associated medical burdens (i.e., cardiometabolic and neurocognitive impairments) have been rising over the past several decades globally. The combination of exercise and ketone supplementation has been recently proposed as one of the solutions with potential clinical value, of which the interventional effects and underlying mechanisms remain unclear. The current study aims at (1) investigating the additive effects of ketone ester supplements to exercise in aspects of cardiorespiratory fitness, metabolism, and neurocognitive status, and (2) examining how the exercise type (HIIE [high-intensity interval exercise] vs. MICE [moderate-intensity continuous exercise]) influences the cardiometabolic and neurocognitive responses of the exercise-diet regime. For each of the 30 participants, six experimental trials will be performed in a randomized trial with a counterbalanced order: (1) HIIE-KT condition (HIIE with ketone supplements); (2) MICE-KT condition (MICE with ketone supplements); (3) NE-KT condition (non-exercise with ketone supplements); (4) HIIE-PLA condition (HIIE with taste-matched placebo); (5) MICE-PLA condition; and (6) NE-PLA condition. Cardiometabolic and neurocognitive parameters will be assessed before and after 30, 60, and 90 min subsequently ketone ester supplements.

ELIGIBILITY:
Inclusion Criteria:

* body mass index > 25 kg/m^2;
* right-handed.

Exclusion Criteria:

* psychiatric, neurologic, cardiovascular, or metabolic disease, including type 1 and type 2 diabetes mellitus;
* addicts to alcohol, nicotine, or drugs;
* oral contraceptive or any medication intake during the past 6 months;
* current engagement in any resistant exercise.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake | 2 weeks
  The measurement name is "maximal oxygen uptake". It will be assessed by cardiopulmonary exercise testing (CPET) equipment, such as cycle ergometers, along with a metabolic cart for measuring oxygen consumption. The unit of measurement is milliliters of oxygen per kilogram per minute(mL/kg/min).
Systolic Blood Pressure | 6 weeks
  The measurement name is "systolic blood pressure". It will be assessed by a blood pressure monitor in laboratory settings. The unit of measurement is millimeters of mercury (mmHg).
Diastolic Blood Pressure | 6 weeks
  The measurement name is "diastolic blood pressure". It will be assessed by a blood pressure monitor in laboratory settings. The unit of measurement is millimeters of mercury (mmHg).
Concentration of Blood Lipid | 6 weeks
  The measurement name is "blood lipid". It will be assessed by the cholestene system in laboratory settings. The unit of measurement is milligrams per deciliter (mg/dL).
Concentration of Blood Glucose | 6 weeks
  The measurement name is "blood glucose". It will be assessed by a glucometer in laboratory settings. The unit of measurement is millimoles per liter (mmol/L).
Concentration of Blood Beta-Hydroxybutyrate | 6 weeks
  The measurement name is "blood beta-hydroxybutyrate". It will be assessed by specific ketone meters designed for beta-hydroxybutyrate measurement. The unit of measurement is millimoles per liter (mmol/L).
Concentration of Blood Lactic Acid | 6 weeks
  The measurement name is "blood lactic acid". It will be assessed by lactate monitor in laboratory settings. The unit of measurement is millimoles per litre (mmol/L).
Concentration of Blood Insulin | 6 weeks
  The measurement name is "blood insulin". It will be assessed by immunoassay system (chemiluminescence immunoassay analyzer) using blood samples. The unit of measurement is microunits per milliliter (μU/mL).
Reaction Time of Stroop Task | 6 weeks
  The measurement name is "reaction time of stroop task". The measurement will be assessed by psychological paradigm named Stroop Task. The unit of measurement is milliseconds (ms).
Accuracy of Stroop Task | 6 weeks
  The measurement name is "accuracy of Stroop task". The measurement will be assessed by psychological paradigm named Stroop Task. Accuracy is generally measured as a percentage (%).
Reaction Time of N-back Task | 6 weeks
  The measurement name is "reaction time of N-back task". The measurement will be assessed by psychological paradigm named N-back task. The unit of measurement is milliseconds (ms).
Accuracy of N-back Task | 6 weeks
  The measurement name is "accuracy of N-back task". The measurement will be assessed by psychological paradigm named N-back task. Accuracy is generally measured as a percentage (%).
Cerebral Hemoglobin Concentration | 6 weeks
  The measurement name is "cerebral hemoglobin concentration". The measurement will be assessed by functional near-infrared spectroscopy (fNIRS). The unit of measurement is micromoles per liter (μM).

SECONDARY OUTCOMES:
Arousal Level | 6 weeks
  The measurement name is "arousal level". It will be assessed by the Two-Dimensional Mood Scale in laboratory settings. The level is scored 0-5 (no special unit).

CONTACTS AND LOCATIONS:
Overall Officials: Zhaowei Kong, PhD, Principal Investigator — University of Macau

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared 2 years after completion. The data will be available for 2 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01/04/2025 - 01/04/2027
Access Criteria: Acquire by request.

REFERENCES:
- [Background] Walsh JJ, Caldwell HG, Neudorf H, Ainslie PN, Little JP. Short-term ketone monoester supplementation improves cerebral blood flow and cognition in obesity: A randomized cross-over trial. J Physiol. 2021 Nov;599(21):4763-4778. doi: 10.1113/JP281988. Epub 2021 Oct 4. PMID 34605026
- [Background] Margolis LM, O'Fallon KS. Utility of Ketone Supplementation to Enhance Physical Performance: A Systematic Review. Adv Nutr. 2020 Mar 1;11(2):412-419. doi: 10.1093/advances/nmz104. PMID 31586177
- [Background] Valenzuela PL, Castillo-Garcia A, Morales JS, Lucia A. Perspective: Ketone Supplementation in Sports-Does It Work? Adv Nutr. 2021 Mar 31;12(2):305-315. doi: 10.1093/advances/nmaa130. PMID 33094332
- [Background] Kesl SL, Poff AM, Ward NP, Fiorelli TN, Ari C, Van Putten AJ, Sherwood JW, Arnold P, D'Agostino DP. Effects of exogenous ketone supplementation on blood ketone, glucose, triglyceride, and lipoprotein levels in Sprague-Dawley rats. Nutr Metab (Lond). 2016 Feb 4;13:9. doi: 10.1186/s12986-016-0069-y. eCollection 2016. PMID 26855664
- [Background] Zhang Y, Kuang Y, LaManna JC, Puchowicz MA. Contribution of brain glucose and ketone bodies to oxidative metabolism. Adv Exp Med Biol. 2013;765:365-370. doi: 10.1007/978-1-4614-4989-8_51. PMID 22879057